CLINICAL TRIAL: NCT06205420
Title: Injection Molding Technique: a Minimally Invasive Management for Enamel Hypoplasia Affecting Permanent Anterior Teeth in Children a Randomized Clinical Trial
Brief Title: Injection Molding Technique: a Minimally Invasive Management for Enamel Hypoplasia Affecting Permanent Anterior Teeth in Children
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Nour Wahba, Lecturer of Pediatric Dentistry, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FDASU-RecIR012365
Record Dates: First submitted 2023-12-05; First posted 2024-01-16 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Enamel Hypoplasia
Keywords: composite resin restoration; giomer; injectable restorations; injection molding; developmental enamel defects; Permanent Anterior teeth
MeSH Terms: conditions — Dental Enamel Hypoplasia; Developmental Defects of Enamel

STUDY DESIGN:
Intervention Model Description: This treatment involves the use of two different injectable restorations for the esthetic treatment of hypoplastic anterior teeth.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Injectable composite resin restoration (Experimental): The use of injectable GC Gaenial restoration in restoring hypoplastic permanent anterior teeth and the evaluation of its clinical performance using FDI criteria.
  Interventions: Drug: Injectable composite resin restoration
- Injectable Giomer restoration (Experimental): The use injectable beautiful flow giomer restoration in restoring hypoplastic permanent anterior teeth and the evaluation of its clinical performance using FDI criteria.
  Interventions: Drug: Injectable giomer restoration

INTERVENTIONS:
Drug: Injectable composite resin restoration — The teeth affected with enamel hypoplasia will be prepared by removing all defective enamel to place the restorations on sound tooth structure as recommended by the IAPD.
  A tooth-by-tooth approach will be employed, where adjacent teeth will be isolated with Teflon tape before selective enamel etching. Selective etching of cut enamel will be done for 15 seconds using 37% phosphoric acid gel. Self-etch adhesive system will be used and highly filled flowable composite will be injected in the accurately positioned transparent clear stent through the small channels created by the tip of the restoration syringe in the incisal edge to restore the affected teeth.
  Curing will be done on the incisal and labial aspects for 20 seconds and will be repeated after clear stent removal for additional 20 seconds. After removal of the clear stent from the patient's mouth, the restoration sprue as well as excess polymerized restoration will be scrapped off with a scalpel.
  Arms: Injectable composite resin restoration
Drug: Injectable giomer restoration — The teeth affected with enamel hypoplasia will be prepared by removing all defective enamel to place the restorations on sound tooth structure as recommended by the IAPD.
  A tooth-by-tooth approach will be employed, where adjacent teeth will be isolated with Teflon tape before selective enamel etching. Selective etching of cut enamel will be done for 15 seconds using 37% phosphoric acid gel. Self-etch adhesive system will be used and an injectable giomer restoration will be injected in the accurately positioned transparent clear stent through the small channels created by the tip of the restoration syringe in the incisal edge to restore the affected teeth.
  Curing will be done on the incisal and labial aspects for 20 seconds and will be repeated after clear stent removal for additional 20 seconds. After removal of the clear stent from the patient's mouth, the restoration sprue as well as excess polymerized restoration will be scrapped off with a scalpel.
  Arms: Injectable Giomer restoration

SUMMARY:
This study aims to evaluate and compare the clinical performance of the injectable giomer restoration versus an injectable composite resin restoration using the injection molding technique for veneering hypoplastic permanent maxillary and mandibular anterior teeth using the FDI criteria. Follow up will be done every 6 months for 2 years.

DETAILED DESCRIPTION:
The aim of this study is to evaluate and compare the two-year clinical performance of injectable giomer restoration to an injectable composite resin restoration using the injection molding technique for veneering permanent maxillary and mandibular anterior teeth affected with enamel hypoplasia in children using the FDI criteria.

Injection molding technique using injectable composite resin restoration and injectable giomer restoration will be implemented for the esthetic management of permanent anterior teeth affected with enamel hypoplasia in children after removal of the defective enamel, its etching and bonding. Evaluation of their performance will be done using FDI criteria and will be followed up for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Healthy patients: Class I according to the American Society of Anaesthesiologists (ASA class I).
* Teeth scored code 3 according to Modified Developmental Defects of enamel (mDDE) index.
* Maxillary and mandibular permanent anterior teeth

Exclusion Criteria:

* Refusal of the parents to sign the informed consent.
* Signs and symptoms of reversible or irreversible pulpitis, as well as necrosis affecting the permanent anterior teeth.
* Enamel hypomineralization

Ages: 8 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 14 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Clinical performance using World Dental Federation (FDI) criteria for evaluating direct restorations. | every 6months for 2 years
  Clinical performance of an injectable giomer compared to composite restoration in permanent anterior teeth with enamel hypoplasia evaluated by FDI criteria to assess the quality of direct restorations. These are divided into functional, biological, esthetic, and miscellaneous properties. The functional properties assess the fracture of material, its retention, the marginal adaptation, the proximal contact point, the form and contour, the occlusion and wear of dental restorations. The biological assess the presence of recurrent caries, the hard dental tissue defect at the restoration margin, postoperative hypersensitivity and pulpal status, while the esthetic evaluates surface luster and texture, marginal staining, and color match. The miscellaneous examines the patient's perspective of the restoration and the radiographic appearance of the restorations. Every domain assessed is given a score from 1-5, where 1 indicates a clinically excellent property and 5 a clinically poor property.

SECONDARY OUTCOMES:
The Mean Annual Failure rate using the World Dental Federation (FDI) criteria. | 1 year
  Calculate the mean annual failure rate or the normalized failure index of the injectable giomer restoration versus the injectable composite resin restoration using the injection molding technique via the FDI criteria. This can be done by several ways: 1) dividing the total failure rate by the number of observation years, 2) using different mathematical formulas given by the FDI for its measurement.
Measuring the impact of enamel hypoplasia on children's daily life from children's and parents' perspectives | 6 months
  Evaluate the impact of enamel hypoplasia on children's life by assessing the oral-health-related quality of life of the treated children before and after treatment using the parental perception, family impact scale questionnaires (P-CPQ and FIS) and child perception questionnaire (CPQ-8-10/ 11-14). The former assess the oral symptoms, functional limitation, and social wellbeing of children from their parents' perspectives and the impact their teeth have on the families' daily life, while the latter assesses the same domains but from the children's perspectives. These are scored from 0-4 according to the answers given by the children and parents, where 0 indicates that 'never', 1 'once or twice', 2 'sometimes', 3 'often' and 4 'every day'. Measuring these questionnaires before and after treatment shows the effect of treatment on their quality of life. A total score is gathered for each domain in the questionnaire and is compared to the scores obtained after 6 months.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry Ain Shams University, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No